CLINICAL TRIAL: NCT02898623
Title: Performances of Immunoassays Based on the Detection of Antibodies Directed Against Mycobacterium Tuberculosis Antigen for the Diagnosis of Active Tuberculosis in Adults
Brief Title: Serological Test for the Diagnosis of TB
Acronym: MycoTB
Status: Terminated | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 9179
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Active Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — Evaluation of performance of immunoassays based on the detection of antibodies directed against Mycobacterium tuberculosis antigen

SUMMARY:
TB remains a health problem in France with about 5,000 new cases per year. Development of new screening tests is a priority for TB. The main objective of the study is to evaluate performances of innovative blood tests to identify active tuberculosis in adults patients living in low-prevalence country. Adult patients with possible TB from will be tested for the presence of antibodies directed against M. tuberculosis selected antigens. Positive and negative predictive values will be established based on TB culture results.

ELIGIBILITY:
Inclusion Criteria:

* Signs of possible Tuberculosis (TB); testing for TB in routine practice (microbiology)

Exclusion Criteria:

* Immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active tuberculosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-12-20 (Actual); Primary Completion 2014-12-20 (Actual); Study Completion 2015-06-20 (Actual)

PRIMARY OUTCOMES:
Positive and negative predictive values for the diagnosis of active TB | 48 months

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Tuaillon, MD; PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital Montpellier Department of microbiology, Montpellier, France

IPD SHARING:
Plan to Share IPD: No